CLINICAL TRIAL: NCT03277755
Title: An Open-label Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Odalasvir and AL-335 Alone and in Combination With Simeprevir in Subjects With Moderately Impaired Hepatic Function
Brief Title: A Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Odalasvir and AL-335 Alone and in Combination With Simeprevir in Participants With Moderately Impaired Hepatic Function
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Development program of JNJ-4178 was discontinued.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108294; 64294178HPC1020 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — adafosbuvir; Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort1:Participants With Moderately Impaired Hepatic Function (Experimental): Participants With moderately impaired hepatic function will receive a single oral dose of AL-335 800 milligram (mg) (2 tablets of 400 mg AL-335) on Day 1 of Part 1 followed by a single oral dose of odalasvir (ODV) 25 mg (1 tablet of 25 mg ODV) on Day 8 of Part 1 and a combination of AL-335 800 mg (2 tablets of 400 mg AL-335) + ODV 25 mg (1 tablet of 25 mg ODV) + simeprevir (SMV) 75 mg (1 capsule of 75 mg SMV) once daily on Day 1 to 14 of Part 2. There will be a washout period between Part 1 and Part 2 of at least 14 days. Day 8 of Part 1 will be the start of the washout period. Prior to the start of study drug administration in Part 2, a safety review will be performed by the Sponsor.
  Interventions: Drug: AL-335 800 mg; Drug: ODV 25 mg; Drug: SMV 75 mg
- Cohort 2: Participants With Normal Hepatic Function (Experimental): Participants with normal hepatic function will receive a single oral dose of AL-335 800 mg (2 tablets of 400 mg AL-335) on Day 1 of Part 1 followed by a single oral dose of ODV 25 mg (1 tablet of 25 mg ODV) on Day 8 of Part 1 and a combination of AL-335 800 mg (2 tablets of 400 mg AL-335) + ODV 25 mg (1 tablet of 25 mg ODV) + SMV 75 mg (1 capsule of 75 mg SMV) once daily on Day 1 to 14 of Part 2. There will be a washout period between Part 1 and Part 2 of at least 14 days. Day 8 of Part 1 will be the start of the washout period. Prior to the start of study drug administration in Part 2, a safety review will be performed by the Sponsor.
  Interventions: Drug: AL-335 800 mg; Drug: ODV 25 mg; Drug: SMV 75 mg

INTERVENTIONS:
Drug: AL-335 800 mg — Participants will receive AL-335 800 mg (2 tablets of 400 mg AL-335) single oral dose on Day 1 of part 1 and in combination as AL-335 + ODV + SMV once daily orally from Day 1 to 14 of part 2.
  Other Names: JNJ-64146212
Drug: ODV 25 mg — Participants will receive ODV 25 mg (1 tablet of 25 mg ODV) single oral dose on Day 8 of part 1 and in combination as AL-335 + ODV + SMV once daily orally from Day 1 to 14 of part 2.
  Other Names: JNJ-64289901
Drug: SMV 75 mg — Participants will receive SMV 75 mg in combination as AL-335 + ODV + SMV once daily orally from Day 1 to 14 of part 2.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of AL-335, odalasvir (ODV) and its metabolites ALS-022399 and ALS-022227, after a single oral dose of ODV and AL-335 respectively, in participants with moderately impaired hepatic function compared to participants with normal hepatic function. Also to evaluate the steady-state PK of AL-335 and its metabolites ALS-022399 and ALS-022227, ODV and simeprevir (SMV) after multiple oral doses of the combination of AL-335+ODV+SMV, in participants with moderately impaired hepatic function compared to participants with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index (BMI; weight in kilogram (kg) divided by the square of height in meters) of 18.0 to 35.0 kilogram per meter square (kg/m^2) extremes included, and a body weight not less than 50.0 kg
* Participant must have a normal 12-lead electrocardiogram (ECG) (based on the mean value of triplicate ECG parameters) consistent with normal cardiac conduction and function at screening, as defined in the protocol
* Absence of findings indicative of hepatocellular carcinoma in an ultrasonography determined within 90 days prior to screening (or between screening and Day -1 of Part 1 of the study)
* Contraceptive use by women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies; a female participant with non childbearing potential must be; a) postmenopausal, or b) surgically sterile. Participant of childbearing potential must; a) have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) pregnancy test at screening and a negative urine beta hCG pregnancy test at baseline (Day -1), and b) not get pregnant from screening until at least 60 days after the end of treatment by adhering to one of the acceptable methods of birth control to avoid pregnancy
* Contraceptive use by men should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies: A male participant: a) must either be surgically sterile, or b) must not be heterosexually active from baseline until at least 60 days after the end of treatment or c) must be practicing an acceptable method of birth control from baseline until at least 60 days after the end of treatment, if heterosexually active with a woman of childbearing potential
* Participants with moderately impaired hepatic function (Cohort 1) must meet the following additional inclusion criteria:

  1. Participants must have a stable hepatic function as confirmed by serum bilirubin, serum albumin, prothrombin, ascites, and hepatic encephalopathy status measured during screening and those measured within 24 hours prior to first study drug administration on Day 1 in Part 1
  2. Participants must be hepatically impaired with a Class B classification as defined by the Child Pugh classification of severity of liver disease, that is, a total Child-Pugh score of 7 to 9, inclusive.
* Participants with normal hepatic function (Cohort 2) must meet the additional inclusion criteria to be enrolled in the study: Participants must have a normal hepatic function as confirmed by serum bilirubin, serum albumin, prothrombin, ascites, and hepatic encephalopathy status measured during screening and those measured within 24 hours prior to first study drug administration on Day 1 in Part 1

Exclusion Criteria:

* Participant has either: a history of renal insufficiency (estimated creatinine clearance lesser than (<) 90 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) for estimated glomerular filtration rate [eGFR] according to the Chronic Kidney Disease Epidemiology Collaboration [CKD- EPI] equation) 18, or serum creatinine grade 1 or greater than (>) 1.1* upper limit of normal [ULN]) during screening
* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (example, compromise the well-being), or that could prevent, limit, or confound the protocol-specified assessments
* Participant with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, or urticarial
* Participant has known allergies, hypersensitivity, or intolerance to simeprevir (SMV), odalasvir (ODV), or AL 335, or their excipients
* Participant who smokes more than 10 cigarettes or 2 cigars or 2 pipes per day from within 90 days before screening until the end of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-11 (Estimated); Primary Completion 2017-12-22 (Estimated); Study Completion 2017-12-22 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentration (Cmax) of AL-335 and its Metabolites ALS-022399 and ALS-022227 | Day 1: Predose, at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours postdose
  Cmax is defined as maximum observed plasma concentration of AL-335 and its metabolites ALS-022399 and ALS-022227.
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC [0-last]) of AL-335 and its Metabolites ALS-022399 and ALS-022227 | Day 1: Predose, at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of AL-335 and its Metabolites ALS-022399 and ALS-022227 | Day 1: Predose, at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 28, 32, 36, 48, 60, and 72 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C (last)/ lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to the time of the last measurable concentration, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Part 1: Maximum Observed Plasma Concentration (Cmax) of Odalasvir (ODV) | Day 8: Predose, at 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  Cmax is defined as maximum observed plasma concentration of ODV.
Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Measurable Concentration (AUC [0-last]) of ODV | Day 8: Predose, at 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ODV | Day 8: Predose, at 1, 3, 4, 5, 6, 7, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, and 168 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C (last)/lambda(z); wherein AUC (last) is area under the plasma concentration-time curve from time zero to the time of the last measurable concentration, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Part 2: Maximum Observed Plasma Concentration (Cmax) of Simeprevir (SMV) | Day 14: Predose, 1, 2, 4, 6, 8, 10, 12, 16 and 24 hours postdose
  Cmax is defined as maximum observed plasma concentration of SMV.
Part 2: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC[0-24]) of SMV | Day 14: Predose, 1, 2, 4, 6, 8, 10, 12, 16 and 24 hours postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours postdose, calculated by linear-linear trapezoidal summation.
Part 2: Maximum Observed Plasma Concentration (Cmax) of ODV | Day 14: Predose, 1, 3, 4, 5, 6, 7, 8, 12, 16 and 24 postdose
  Cmax is defined as maximum observed plasma concentration of ODV.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours Postdose (AUC[0-24]) of ODV | Day 14: Predose, 1, 3, 4, 5, 6, 7, 8, 12, 16 and 24 postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours postdose, calculated by linear-linear trapezoidal summation.
Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of ODV | Day 14: Predose, 1, 3, 4, 5, 6, 7, 8, 12, 16 and 24 postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C (last)/ lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Part 2: Maximum Observed Plasma Concentration (Cmax) of AL-335 and its Metabolites ALS-022399 and ALS-022227 | Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours postdose
  Cmax is defined as maximum observed plasma concentration of AL-335 and its metabolites ALS-022399 and ALS-022227.
Part 2: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours (AUC[0-24]) Postdose of AL-335 and its metabolites ALS-022399 and ALS-022227 | Day 14: Predose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours postdose
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours postdose, calculated by linear-linear trapezoidal summation.

SECONDARY OUTCOMES:
Part 1 and 2: Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to 30-35 days after last drug intake (approximately up to 102 days)
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC